CLINICAL TRIAL: NCT06255223
Title: An Open-label, Single-arm Study to Evaluate the Efficacy and Safety of Multimodal Radiotherapy in the Treatment of Renal Cell Carcinoma Progressed After Prior Immunotherapy
Brief Title: A Study of Multimodal Radiotherapy for Renal Cell Carcinoma Progressed After Prior Immunotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Le Qu, Associate chief urologist, Jinling Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024DZKY-018-01
Record Dates: First submitted 2024-02-03; First posted 2024-02-13 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Renal Cell Carcinoma; Radiotherapy; Immune Checkpoint Inhibitor
Keywords: RCC; Multimodal radiotherapy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Radiotherapy; Radiosurgery; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental group (Experimental): For eligible subjects, multimodal radiotherapy will be added to the treatment besides original immunotherapy or combinations of immunotherapy and TKIs after adjustment.
  Interventions: Radiation: High-dose Radiotherapy (HDRT); Radiation: Low-dose Radiotherapy (LDRT); Drug: Anti-PD-1 monoclonal antibody

INTERVENTIONS:
Radiation: High-dose Radiotherapy (HDRT) — SBRT was adopted, and radiotherapy plan was made according to the location and size of lesions (total dose 20-70Gy, 5-12Gy every time).
  Other Names: Stereotactic Body Radiation Therapy; SBRT; Stereotactic Ablative Body Radiation Therapy; SABR
Radiation: Low-dose Radiotherapy (LDRT) — Radiotherapy plan was made according to the location and size of lesions (total dose 2Gy, 1Gy every time). After completing SBRT, LDRT was performed on as many metastatic sites as possible.
Drug: Anti-PD-1 monoclonal antibody — At the end of multimodal radiotherapy, immunotherapy was given within 7 days and in a subsequent LDRT. The maximum duration is 24 months.

SUMMARY:
The objective of this single-center clinical study was to evaluate the disease control rate(DCR) and safety of multimodal radiotherapy in the treatment of patients with renal cell carcinoma (RCC) progressed after prior immunotherapy.

DETAILED DESCRIPTION:
The patients who were clinically diagnosed advanced renal cell carcinoma with progression after 1-2 previous systemic therapies (at least one regimen containing immune checkpoint inhibitors, including combined VEGFR-TKI drugs), with two or more metastases at different sites, will be evaluated by the researchers. For eligible subjects, multimodal radiotherapy will be added to the treatment besides original immunotherapy or combinations of immunotherapy and TKIs after adjustment. The disease control rate and safety of this treatment will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Renal cell carcinoma confirmed histologically or cytopathologically, including unresectable or recurrent metastatic renal cell carcinoma.
* Subject's previous treatment: Disease progression or intolerance following prior treatment with 1-2 systemic therapies (at least one regimen containing immune checkpoint inhibitors, including combined VEGFR-TKI drugs), And patients who have progressed within 12 months of prior immunoadjuvant or neoadjuvant therapy; According to the evaluation of attending physicians and professional radiotherapy doctors, it meets the standard of radiotherapy.
* Patients can tolerate sequential immunotherapy while receiving radiation therapy.
* At least two or more metastases at different sites are considered observable according to RECIST v1.1.
* Subjects have fully understood and voluntarily signed an informed Consent form (ICF).
* ECOG 0-1 points.
* Major organs are functioning well.
* Willing and able to comply with study plan visits, treatment laboratory tests, sample retention, and other procedures.
* Fertile women must voluntarily use a highly effective contraceptive method (e.g., oral, injectable or implantable, barrier method, spermicide and condom, or intrauterine device) from the study period to ≥120 days after the last dose and have negative urine or serum pregnancy test results ≤7 days prior to enrolment.
* Male patients who are not sterilized must voluntarily use highly effective contraception during the study period until ≥120 days after the last dose.

Exclusion Criteria:

* A history of malignancies other than the disease studied within the past 5 years, other than malignancies that are expected to be cured with treatment (including but not limited to adequately treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell skin cancer, or breast ductal carcinoma in situ treated with radical surgery).
* Systemic treatment with other antitumor agents, including targeted agents, immunotherapy agents and their combination regimens (eligible for inclusion after 5 half-lives), local antitumor therapy, or clinical investigational drug or device therapy, was administered 4 weeks prior to the first study.
* Previous history of radiation therapy at any site or in any mode.
* Had major surgery (as judged by the investigator) within 4 weeks prior to the first trial or was convalescing.
* A history of severe drug allergy, including but not limited to antibody drugs.
* Patients with contraindications to restart immunotherapy.
* A known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation may require long-term adrenal corticosteroid therapy.
* Patients with thyroid, suprarenal, or hypopituitarism that can be controlled with hormone replacement therapy alone, type 1 diabetes, and psoriasis or vitiligo that do not require systemic treatment are eligible to participate in this study.
* Toxicity did not resolve after previous antitumor therapy, i.e. regression to baseline, prescribed grade 0 to 1 (except alopecia) as defined in NCI-CTCAE 5.0, or to the levels specified in the inclusion/exclusion criteria. Irreversible toxicity (such as hearing loss) that could reasonably be expected not to be aggravated by the drug under study could be included in this study.
* Have central nervous system metastases and/or cancerous meningitis.
* A known history of clinically significant liver disease.
* Accompanied by uncontrolled third space effusion requiring repeated drainage, such as pleural effusion, ascites, pericardial effusion, etc.
* In the first study, systemic corticosteroids or other immunosuppressive drugs were administered within 14 days prior to medication.
* Patients with any severe or uncontrolled disease.
* Have or have a suspected presence of active autoimmune diseases, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, etc.
* Renal failure requires hemodialysis or peritoneal dialysis.
* A history of immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation.
* History of live attenuated vaccine vaccination within 4 weeks prior to administration or expected live attenuated vaccine vaccination during the study period was studied for the first time.
* People who have a history of psychotropic substance abuse and cannot abstain or have a history of mental disorders.
* Pregnant or lactating women.
* Other severe, acute, or chronic medical or psychiatric conditions or laboratory abnormalities, as determined by the investigator, that may increase the risks associated with study participation or that may interfere with the interpretation of the study results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR) | Up to 1 year
  After completing the full course of radiotherapy, the patients underwent periodic imaging evaluation. Tumor imaging evaluations within 48 weeks should be performed every 6 weeks (±7 days) and every 12 weeks (±7 days) after 48 weeks until disease progression, loss of follow-up, death, withdrawal of study informed consent, subject initiation of other antitumor therapy, or study termination. DCR was evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST v 1.1).
Incidence of adverse events | Up to 1 year
  Adverse events according to Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0). The patients must be on the trial for at least 8 weeks. Adverse events must be attributable to radiation therapy or immunotherapy.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 1 year
  After completing the full course of radiotherapy, the patients underwent periodic imaging evaluation. Tumor imaging evaluations within 48 weeks should be performed every 6 weeks (±7 days) and every 12 weeks (±7 days) after 48 weeks until disease progression, loss of follow-up, death, withdrawal of study informed consent, subject initiation of other antitumor therapy, or study termination. PFS was evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST v 1.1).
Objective response rate (ORR) (partial response or complete response) | Up to 1 year
  After completing the full course of radiotherapy, the patients underwent periodic imaging evaluation. Tumor imaging evaluations within 48 weeks should be performed every 6 weeks (±7 days) and every 12 weeks (±7 days) after 48 weeks until disease progression, loss of follow-up, death, withdrawal of study informed consent, subject initiation of other antitumor therapy, or study termination. ORR was evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST v 1.1).
Overall survival (OS) | Up to 1 year
  After completing the full course of radiotherapy, patients were followed for one year until the last visit or death. OS was measured based on data collected through professional procedures.
Abscopal effects | 1 year
  When making a radiotherapy plan, identify one or more LDRT lesions to be used for puncture. After the completion of the full course of radiotherapy, the predetermined lesions were punctured, and the obtained specimens were analyzed by pathological biopsy and immunohistochemistry to evaluate the changes of tumor microenvironment. At the same time, the patient's blood was extracted and the relevant cytokines were detected for analysis.
Change of lymphocyte subsets and tumor-associated macrophages (TAMs) | 1 year
  When making a radiotherapy plan, identify one or more LDRT lesions to be used for puncture. After the completion of the full course of radiotherapy, the predetermined lesions were punctured, and the obtained specimens were analyzed by pathological biopsy and immunohistochemistry to evaluate the changes of immune cells through the markers in tumor microenvironment. At the same time, the patient's blood was extracted and the numbers of relevant cells were detected. The changes of CD8+ T cells, CD4+ T cells, Treg, phenotype of TAMs and DCs were evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling Hospital, Affiliated Hospital of Medical School, Nanjing University, Nanjing, Jiangsu, China